CLINICAL TRIAL: NCT05281354
Title: Development of a Personalised Therapeutic Approach for Cancer Patients With Resting Hypermetabolism
Acronym: METABO-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHM-2021/S13/12
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-03

CONDITIONS: Cancer
Keywords: Hypermetabolism; Rest Energy Expenditure; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (No Intervention): Follow-up according to standard practice
- multimodal intervention (Experimental): Addition of a treatment to normalise resting energy expenditure according to the observed abnormalities
  Interventions: Other: Multimodal intervention

INTERVENTIONS:
Other: Multimodal intervention — Treatment to normalise resting energy expenditure according to the observed abnormalities such as anti-inflammatory treatment with Omega 3 in the case of systemic inflammation, treatment with a non-specific beta-blocker such as propanolol in the case of activation of the beta-adrenergic system, appropriate physical activity in the case of sarcopenia, or nutritional support aimed at re-establishing the balance of calorie and protein intake and expenditure, or a combination of these actions
  Arms: multimodal intervention

SUMMARY:
Half of all cancer patients show an increase in resting energy expenditure. The causes of hypermetabolism have only recently been investigated in cancerology. One established cause is inflammation, but other causes have yet to be identified.

The interest in hypermetabolism is due to the fact that it appears early, before the onset of clinical deterioration (weight loss, sarcopenia, altered performance status) and that it correlates with patient morbidity and mortality. Like the other parameters that make up cachexia, it is both a predictor of toxicity and reduced efficacy of anti-tumour treatments and a prognostic factor, regardless of the tumour.

A therapeutic goal is to correct hypermetabolism for two reasons:

* avoid progression to clinical cachexia, which is an independent cause of morbidity and mortality
* increase the efficacy of anti-PD1/PDL1 immunotherapies. This new class of therapy has revolutionised the therapeutic management of many cancers but is less effective in cases of inflammation and/or altered performance status and/or hypermetabolism.

Investigator hypothesises that it is possible to develop a patient-specific treatment to correct hypermetabolism, depending on the predominant clinical or biological cause.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with solid malignancy (any possible primary tumor), stage IV (M1), progressive or stable
* Without treatment or with anti-tumour treatment
* WHO performance status ≤ 2
* Person affiliated or benefiting from a social security scheme
* Having signed a consent to participate in the study
* Patient with hypermetabolism at the inclusion visit

Exclusion Criteria:

* Patient agitated, or unable to understand or tolerate wearing a mask for 20 minutes
* No active tumour disease (complete remission or ongoing tumour response)
* Care plan that does not allow for two calorimetry sessions 1 month apart
* Pregnant, breastfeeding or parturient woman
* Person deprived of liberty by judicial or administrative decision
* Person subject to forced psychiatric care
* Person subject to a legal protection measure
* Inclusion in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Assess the impact at 1 month of a multimodal intervention on hypermetabolism in cancer patients compared to standard care | 1 month after inclusion
  The impact of a multimodal intervention is evaluated by proportion of hypermetabolic patients at 1 month in the personalised multimodal intervention arm compared to patients in the standard care arm

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Du Mans, Le Mans
  - Hôpital COCHIN, Paris